CLINICAL TRIAL: NCT05384353
Title: In Vivo PET of Synaptic Density in Cognitive Disorders: Prospective Evaluation of Neuronal Dysfunction and Relation to Symptomatology
Brief Title: In Vivo PET of Synaptic Density in Cognitive Disorders
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S66111; 2021-006610-36 (EudraCT Number)
Record Dates: First submitted 2022-04-06; First posted 2022-05-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Frontotemporal Degeneration; Dementia With Lewy Bodies; Psychiatric Disorder
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Mental Disorders | interventions — SynVesT-1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy controls: Synaptic density PET-MR and neuropsychological testing
  Interventions: Other: [18F]-SynVesT-1
- Patients with Alzheimer's disease: Synaptic density PET-MR and additional neuropsychological testing (if necessary)
  Interventions: Other: [18F]-SynVesT-1
- Patients with Frontotemporal degeneration: Synaptic density PET-MR and additional neuropsychological testing (if necessary)
  Interventions: Other: [18F]-SynVesT-1
- Patients with Dementia with Lewy Bodies: Synaptic density PET-MR and additional neuropsychological testing (if necessary)
  Interventions: Other: [18F]-SynVesT-1
- Patients with late-life psychiatric disorders: Synaptic density PET-MR and additional neuropsychological testing (if necessary)
  Interventions: Other: [18F]-SynVesT-1

INTERVENTIONS:
Other: [18F]-SynVesT-1 — PET radioligand binding to synaptic vesicle protein 2A as a proxy for synaptic density

SUMMARY:
This study will compare the discriminative power of [18F]-SynVesT-1 PET and the standard-of-care [18F]-FDG PET in different cognitive disorders (Alzheimer's disease, Frontotemporal degeneration, dementia with Lewy bodies and late-life psychiatric disorders). Moreover, changes in [18F]-SynVesT-1 PET will be evaluated as well as their correlation with specific symptomatology.

DETAILED DESCRIPTION:
Forty healthy controls will be included as well as 110 patients that were referred by the UZ Leuven memory clinic with uncertain diagnosis of cognitive impairment and are already sent for [18F]-FDG PET imaging in their workup (estimated subgroup size: 30 patients with final diagnosis AD (aMCI); 20 patients with DLB; 30 patients with FTD; 30 patients with late-life psychiatric disorder).

Scans will be acquired on a 3T GE Signa PET-MR scanner, for 90 minutes starting at injection of 150 MBq [18F]-SynVesT-1 for healthy controls, and from 60 to 90 minutes post injection of 150 MBq [18F]-SynVesT-1 for patients. For healthy controls, discrete arterial blood samples will be manually collected every 10s from 10 to 90s; every 15s from 90s to 3min; and then at 3.5, 5, 6.5, 8, 12, 15, 20, 25, 30, 45, 60, 75 and 90min. Plasma samples for correction of radiometabolites will be collected at 3, 8, 15, 30, 60 and 90min after injection.

All healthy controls will also be subjected to a neuropsychological test battery and if necessary, additional limited neuropsychological testing on top of those from the memory clinic will be carried out in patients.

ELIGIBILITY:
1. Healthy controls:

   Inclusion Criteria:
   * Age between 18 and 85 years old (aimed to be evenly spread over age intervals).
   * Subject is judged to be in good health by the investigator on the basis of medical history, physical examination including vital signs, clinical laboratory test and urinalysis.
   * No history or evidence of current major neurological, internal or psychiatric disorder, based on the medical assessment and neuropsychological assessment.
   * In subjects < 60 years of age, an unremarkable structural MRI scan as assessed by expert radiologist. In subjects >= 60 years of age white matter hyperintensities corresponding to a white matter lesion (WML) score <= 2 (of 3) on the Age-Related White Matter changes scale are acceptable.
   * When older than 50 years of age, subject is willing to undergo an additional 18F-NAV-4694 scan when cerebral amyloid status is unknown.

   Exclusion Criteria:
   * Subject has a history of any major disease that may interfere with the investigations or make the subject unfit for participation according to the interpretation by the investigator (especially liver and kidney disease, uncontrolled diabetes or most forms of cancer).
   * Subject has any history of a major neurological disorder or known cerebral structural abnormalities.
   * Subject is first-degree relative (sibling, parent or children) of a person with neurological or psychiatric history assessed by a neurologist or psychiatrist (in particular dementia).
   * Evidence of cognitive impairment as assessed by a MMSE score < 28.
   * Subject has a history or evidence of psychiatric disease, as assessed by a validated psychiatric symptom self-assessment tool (Symptom Checklist-90, Beck Depression Inventory (BDI) and Geriatric Depression Scale (GDS)).
   * Subject is currently a user (including ''recreational use'') of any illicit drugs, including cannabis, or has a history of drug or alcohol abuse.
   * Subject chronically uses medication that has central nervous system effects (e.g., opioids, neuroleptics, sedatives, anti-depressants, sleep medication).
   * Subject has had exposure to ionizing radiation (> 1 mSv) in other research studies within the last 12 months.
   * Subject has a contra-indication for MRI scanning.
   * Subject suffers from claustrophobia or cannot tolerate confinement during PET-MRI scanning procedures; subject cannot lie still for approximately 90 minutes inside the scanner.
   * Subject is unwilling to avoid unusual, unaccustomed, or strenuous physical activity (i.e., weightlifting, running, bicycling) from the time of the pre-study visit until the end of scanning.
   * Subject does not understand the study procedures.
   * Subject is unwilling or unable to perform all of the study procedures or is considered unsuitable in any way by the principal investigator.
   * Subject is pregnant (according to Ulti Med hCG urine test) or breastfeeding.
   * Subject is a woman of childbearing potential (WOCBP) who does not agree to apply appropriate contraception methods during study participation and continues to do so for at least 6 months after study completion. For WOCBP: contraception methods with a relatively high Pearl index (natural methods, minipill outside postpartum period, spermicides or condoms in monotherapy or no usage of contraception when sexually active) are not accepted.
   * Subject is a man with a pregnant or non-pregnant WOCBP partner, who does not agree to use a condom and continue to do so until 90 days after study completion. In addition, the non-pregnant WOCBP partner should use a highly effective method of contraception.
   * Subject does not agree that incidental findings are communicated to the general practitioner and to the participant him/herself.
   * Subject is on anticoagulant therapy.
2. Patients:

Inclusion Criteria:

* Patients referred with uncertain diagnosis and subsequent need for FDG PET brain in their work- up to differentiate between dementing disorders or to exclude dementia in late-onset psychiatric disorders with cognitive impairment.
* A routine neuropsychological assessment has been performed during clinical work-up in the memory clinic.
* Subject is at least 30 years old.

Exclusion Criteria:

* Subject has a history or evidence of other major neurological, major psychiatric or major internal pathology that may make him/her unfit for participation according to the interpretation by the investigator (including cardiac, lung, hematological, gastro-intestinal disorders or most forms of cancer).
* Subject's neurological condition has a predominant impact on motor function.
* Subject has no objective cognitive-behavioral deficit based on neuropsychological assessment.
* Subject has important vascular changes abnormal for age or other structural lesions on MR.
* Subject is currently a user (including ''recreational use'') of any illicit drugs, including cannabis, or has a history of drug or alcohol abuse.
* Subject has had exposure to ionizing radiation (> 1 mSv) in other research studies within the last 12 months.
* Subject has a contra-indication for MRI scanning.
* Subject suffers from claustrophobia or cannot tolerate confinement during PET-MRI scanning procedures; subject cannot lie still for 30 minutes inside the scanner.
* Subject is unwilling to avoid unusual, unaccustomed, or strenuous physical activity (i.e., weightlifting, running, bicycling) from the time of the pre-study visit until the end of scanning.
* Subject does not understand the study procedures or does not have a guardian who understands the study procedures.
* Subject (or guardian) is unwilling or unable to perform all of the study procedures or is considered unsuitable in any way by the principal investigator.
* Subject does not agree that incidental findings are communicated to the general practitioner and to the participant him/herself.
* Subject is pregnant (according to Ulti Med hCG urine test) or breastfeeding.
* Subject is a woman of childbearing potential (WOCBP) who does not agree to apply appropriate contraception methods during study participation and continues to do so for at least 6 months after study completion. For WOCBP: contraception methods with a relatively high Pearl index (natural methods, minipill outside postpartum period, spermicides or condoms in monotherapy or no usage of contraception when sexually active) are not accepted.
* Subject is a man with a pregnant or non-pregnant WOCBP partner, who does not agree to use a condom and continue to do so until 90 days after study completion. In addition, the non-pregnant WOCBP partner should use a highly effective method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 healthy controls and 110 patients with uncertain diagnosis of cognitive impairment. All groups should include both sexes. Healthy controls should be evenly spread between the ages of 18 until 85.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Comparison of the discriminative power of [18F]-SynVesT-1 PET and the standard-of-care [18F]-FDG PET in different cognitive disorders | Patients will be included after they underwent [18F]-FDG PET. Estimated time between [18F]-SynVest-1 and [18F]-FDG PET is about 3 months. Estimated visit length for [18F]-SynVest-1 PET is 3 hours. Data analysis will be done when all subjects are scanned.
  Anonymized [18F]-SynVest-1 and [18F]-FDG PET scans from patients with Alzheimer's disease, Frontotemporal degeneration, Dementia with Lewy Bodies or late-life pyschiatric disorders will be evaluated by expert raters blinded to the final diagnosis in order to compare the discriminative power of both tracers.
Synaptic density changes | Neuropsychological evaluation will be performed on the day of the [18F]-SynVesT-1 PET. Estimated visit length is 3 hours. Data analysis will be done when all subjects are scanned.
  [18F]-SynVesT-1 synaptic density changes in different cognitive disorders and correlation with symptomatology

CONTACTS AND LOCATIONS:
Overall Officials: Koen Van Laere, MD, PhD, DSc, Principal Investigator — UZ/KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vanderlinden G, Carron C, Vandenberghe R, Vandenbulcke M, Van Laere K. In vivo PET of synaptic density as potential diagnostic marker for cognitive disorders: prospective comparison with current imaging markers for neuronal dysfunction and relation to symptomatology - study protocol. BMC Med Imaging. 2024 Feb 12;24(1):41. doi: 10.1186/s12880-024-01224-5. PMID 38347458